CLINICAL TRIAL: NCT02063321
Title: Reading Center - Occurence of Diabetic Macular Edema in Patients With Diabetes Mellitus in Slovak Republic
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Emil Martinka (Other)
Collaborators: Novartis Slovakia, s.r.o. (Industry)
Responsible Party: Sponsor-Investigator, Emil Martinka, Head of Diabetology Department, National Institute of Endocrinology and Diabetology, Slovakia
Organization: National Institute of Endocrinology and Diabetology, Slovakia (Other)
Other Study IDs: LUB012013
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-02

CONDITIONS: Diabetic Macular Edema; Diabetic Retinopathy
Keywords: DME, diabetic retinopathy, diabetes mellitus, epidemiology
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of the study is to find out prevalence of diabetic macular edema (DME) in patients with diabetes mellitus in Slovak Republic.The outcome of the project will be epidemiology survey, prevalence of wet form of Diabetic Macular Edema in relation to duration of diabetes, type of diabetes, treatment (insulin vs. OAD or combination) etc. and identification of prognostic factors leading to development of DME.

DETAILED DESCRIPTION:
Epidemiological study, prospective, non-interventional

1. Patient with history of diabetes ≥ 10 years or with suspected visual impairment will be enrolled and screened in NIED during hospitalization
2. Anamnesis and history of diabetes, other co-morbidities, treatment will be recorded
3. Patient undergo in NIED detailed diabetology examination and basic ophthalmology examination (best non-corrected visual acuity in ETDRS score and Amsler grid test)
4. Patient undergo in NIED examination of the back of the eye using fundus camera to take images of retina to assess long-term changes of macula, optic disc, retina vessels and surrounding tissues
5. The assessment of the ophthalmology examination will be carried out in one of two specialized reading centers - II. Eye Clinic SZU FNsP F.D.R., Banská Bystrica or OFTAL Specialized Hospital for Ophthalmology, Zvolen by Retina specialist

The process of screening will be continuous, whilst each patient will sign an informed consent.

Patients records will be stored electronically and data transmission between NIED and Reading Center will be protected using validated and secured software.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years treated in National Institute of Endocrinology and Diabetology
* Patients diagnosed with Diabetes mellitus type I and type 2 respectively
* Presence of Diabetes ≥10 years or patients with suspected visual impairment (duration of diabetes <10 years)
* Signed patient´s information and informed content

Exclusion Criteria:

* Non-compliant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults regularly examined in National Institute of Endocrinology and Diabetology (NIED) for their severity and complications of diabetes will undergo a screening procedure using fundus camera to assess the back of the eye (fundus examination).
Sampling Method: Probability Sample
Enrollment: 762 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Diabetic Macular Edema or clinically significant Diabetic Macular Edema | Patients screened during hospitalization in National Institute of Endocrinology and Diabetology (NIED), usually in 10 days
  Image of fundus taken in NIED securely sent via internet and electronic Clinical Report Form (eCRF) to ophthalmology reading center to assess stage and severity of potential retina damage, feedback to NIED within the stay of screened individual essential for further disease management

SECONDARY OUTCOMES:
Patient´s structure with DME and clinically significant DME in terms of demography and anamnesis of diabetes | Patients screened during hospitalization in NIED, usually in 10 days
Range of visual deterioration and occurence of blindness in relation to duration of diabetes | Patients screened during hospitalization in NIED, usually in 10 days
Prognostic factors, which determine the occurence of DME using explorative analysis | Patients screened during hospitalization in NIED, usually in 10 days
Range of visual deterioration and occurence of blindness in relation to type of diabetes | Patients screened during hospitalization in NIED, usually in 10 days
Range of visual deterioration and occurence of blindness in relation to general treatment (insulin vs. OAD or combination therapy) | Patients screened during hospitalization in NIED, usually in 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Marta Ondrejkova, MD, Study Chair — II. Eye Clinic SZU of F.D.Roosevelt Hospital, Banska Bystrica; Monika Gajdosova, MD, Study Chair — Oftal, s.r.o. Specialized Hospital for Ophthalmology, Zvolen; Emil Martinka, MD, Principal Investigator — Department of Diabetology of National Institute for Endocrinology and Diabetology, Lubochna

REFERENCES:
- See also: Main Site of Principal Investigator — http://www.nedu.sk